CLINICAL TRIAL: NCT07328880
Title: Comparative Study Between Using a 4-L Split-dose Polyethylene Glycol and Bisacodyl + Docusate Sodium Regimen Versus a 2-L Split-dose Polyethylene Glycol Plus Oral Simethicone Regimen Versus Conventional Method for Bowel Preparation Before Colonoscopy
Brief Title: 4-L Split-dose Polyethylene Glycol and Bisacodyl and Docusate Sodium Regimen Versus 2-L Split-dose Polyethylene Glycol Plus Oral Simethicone Regimen for Bowel Preparation Before Colonoscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Rania Mamdouh Elkafoury, Lecturer of Tropical Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 36264PR1193/4/25
Record Dates: First submitted 2025-12-27; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Colonoscopy Preparation
MeSH Terms: interventions — Bisacodyl; Dioctyl Sulfosuccinic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 4-L split-dose polyethylene glycol and Bisacodyl + docusate sodium. (Experimental): 150 patients will be randomized to receive PEG and were instructed to mix four sachets of PEG (Moviprep) in 4 liters of water and drink it over a period of 8 hours starting at 09:00 a.m. and Biscodyl 10 mg + Docusate sodium 100 mg (Minalax) 8 tablets.
  Interventions: Drug: 4-L split-dose polyethylene glycol and Bisacodyl + Docusate sodium.
- 2-L split-dose polyethylene glycol plus oral simethicone regimen . (Active Comparator): 150 patients will be randomized to receive PEG with simethicone and instructed to mix two sachets of PEG (Moviprep) in 2 liters of water and drink it over a period of 4 hours starting at 09:00 a.m. with simethicone (Flatidyl) 4 tablets.
  Interventions: Drug: 2-L split-dose polyethylene glycol plus Oral Simethicone regimen .
- 2-L split-dose polyethylene glycol regimen (control). (Active Comparator): 150 patients will be randomized to receive PEG with simethicone and instructed to mix two sachet of PEG (moviprep) in 2 liters of water and drink it over a period of 4 hours starting at 09:00 a.m.
  Interventions: Drug: 2-L split-dose polyethylene glycol regimen

INTERVENTIONS:
Drug: 4-L split-dose polyethylene glycol and Bisacodyl + Docusate sodium. — Patients who were randomized to receive PEG were instructed to mix four sachets of PEG (Moviprep) in 4 liters of water and drink it over a period of 8 hours starting at 09:00 a.m. and Biscodyl 10 mg + Docusate sodium 100 mg (Minalax) 8 tablets.
  Arms: 4-L split-dose polyethylene glycol and Bisacodyl + docusate sodium.
Drug: 2-L split-dose polyethylene glycol plus Oral Simethicone regimen . — Patients who are randomized to receive PEG with simethicone are instructed to mix two sachets of PEG (Moviprep) in 2 liters of water and drink it over a period of 4 hours starting at 09:00 a.m. with simethicone (Flatidyl) 4 tablets.
  Arms: 2-L split-dose polyethylene glycol plus oral simethicone regimen .
Drug: 2-L split-dose polyethylene glycol regimen — Patients who are randomized to receive PEG with simethicone instructed to mix two sachet of PEG (moviprep) in 2 liters of water and drink it over a period of 4 hours starting at 09:00 a.m.
  Arms: 2-L split-dose polyethylene glycol regimen (control).

SUMMARY:
The goal of this randomized controlled trial is to compare the safety, compliance, and efficacy of different bowel preparation methods prior to colonoscopy. Researchers will compare 4-L split-dose polyethylene glycol and the bisacodyl + docusate sodium regimen versus 2-L split-dose polyethylene glycol plus oral simethicone regimen versus the conventional method for bowel preparation before colonoscopy. Participants will undergo history-taking, clinical examination, laboratory investigations, and colonoscopy. Patients will be randomly assigned to receive 4-L split-dose polyethylene glycol and bisacodyl + docusate sodium, a 2-L split-dose polyethylene glycol regimen plus oral simethicone, or 2-L split-dose polyethylene glycol alone as a control. Colonoscopy will be done 24 hrs after the start of medication. Researchers will assess the quality of the bowel preparation using the Aronchick bowel preparation scale. Researchers will also assess the number of adverse events and ask the patients about the ease of bowel preparation administration, tolerability of preparation regimen, and willingness to take the same agent again for a repeat colonoscopy in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing colonoscopy as a day-care procedure for various indications (lower GI bleeding, colorectal cancer screening, altered bowel habits, etc.)
* Patients of either sex aged >18 years and <70 years.
* Patients willing to give written informed consent.

Exclusion Criteria:

* Presence of Renal failure, cirrhosis, ascites, CCF, bleeding disorders, seizure disorder, gastrointestinal obstruction, or perforation.
* History of serious adverse events to other electrolyte-based colonic lavages.
* Female patients who are pregnant or lactating or considering pregnancy.
* Allergy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-26 (Estimated)

PRIMARY OUTCOMES:
Performing a complete and successful full colonoscopy. | through study completion, an average of 1 year
  Bowel preparation administration, whether completed or not, and the reason for it will be recorded. Assessment of the quality of the bowel preparation using the Aronchick bowel preparation scale.

SECONDARY OUTCOMES:
Bowel preparation side effects | through study completion, an average of 1 year
  Any adverse events (like nausea, vomiting, dizziness, pain abdomen, bloating and anal irritation) will be recorded.
Ease of bowel preparation administration | through study completion, an average of 1 year
  Patients were asked to rate the ease of administration and taste as easy/tolerable/difficult/intolerable.
Tolerability assessment | through study completion, an average of 1 year
  the tolerability is assessed based on whether the patient would take the preparation again in case repeat colonoscopy is required and rate the product as excellent/good/satisfactory/bad.

CONTACTS AND LOCATIONS:
Overall Officials: Nabila A Elgazzar, MD, Study Director — Tropical medicine and infectious diseases Department, Faculty of Medicine, Tanta University
Locations (1):
- Tanta University Hospitals, Tanta, Gharbyea, Egypt